CLINICAL TRIAL: NCT01711268
Title: Correlating Renal Cell Cancer Treatment Efficacy With Sunitinib Therapeutic Levels and Outcomes
Brief Title: Sunitinib Drug Levels and Outcomes in Kidney Cancer
Acronym: CRESTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Howard Gurney, Associate Professor, Western Sydney Local Health District
Other Study IDs: HGWH008
Record Dates: First submitted 2012-08-02; First posted 2012-10-22 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Renal Cell Carcinoma
Keywords: Sunitinib; Renal Cell Carcinoma; Therapeutic Drug Monitoring; Pharmacokinetic; Treatment toxicity
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Sunitinib is an oral drug used for treatment of advanced kidney cancer. The standard dose is 50mg, but many patients require a dose decrease due to side-effects. Drug levels of sunitinib vary approximately 10-fold between patients.

This study will measure blood levels of sunitinib and its metabolite, and correlate these with side-effects and the response to the treatment. The study aims to establish whether blood levels change with time, and see how useful blood levels are for monitoring patients treated with sunitinib.

DETAILED DESCRIPTION:
Rationale: Sunitinib is an oral multi-targeted tyrosine kinase inhibitor used for first-line systemic therapy in metastatic renal cell carcinoma. It is metabolised to a pharmacologically active metabolite, SU012662, which is of equal potency to the parent compound. At a standard 50mg daily dose, variability in plasma levels between patients is approximately ten-fold. In clinical trials, over 30% of patients require a dose reduction due to toxicity. However, some patients can tolerate up to 100mg without excessive toxicity. It is unknown if sunitinib clearance changes with time. Pre-clinical experiments observed tyrosine kinase inhibition at a plasma concentration of 50-100ng/ml.

Design: This is a prospective non-randomized, Phase II clinical study. Decision to treat patients with single-agent sunitinib is pre-determined by treating specialists before entering this study. Toxicity and trough sunitinib/metabolite levels will be measured every six weeks during treatment.

Aim: This study will prospectively examine the relationship between steady-state trough levels of sunitinib/metabolites and the time on treatment, in addition to changes in trough levels over time. Trough levels will also be correlated with other measures of efficacy and treatment-related toxicity. Furthermore, we aim to confirm that the putative target of 50ng/ml correlates with toxicity and time on sunitinib.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal cell cancer treated with single agent sunitinib
* No known primary liver disease and no other severe or uncontrolled concurrent medical conditions
* Signed informed consent

Exclusion Criteria:

* Patients who are unable to sign informed consent
* Patients unable to give blood
* Patients who are pregnant, nursing or not using an effective contraception method
* Patients who had bone-marrow-transplantation prior to sunitinib treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults being treated with sunitinib monotherapy for metastatic renal cell carcinoma
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure (time on sunitinib treatment) | Sunitinib duration (median)
  This duration extends from the date the patient starts sunitinib until the date sunitinib is abandoned. The group with sunitinib concentration below the population median are expected to have a median Time to Treatment Failure (TTF) of approximately 8 months, compared with 14 months in those with sunitinib concentration above the population median.

SECONDARY OUTCOMES:
Toxicity | Every 6 weeks
  Pre-specified toxicities (BP, fatigue, diarrhoea, stomatitis, hand-foot syndrome) will be graded every 6 weeks
Overall survival | 2 years
  Measured from the date of starting sunitinib treatment to the date of death from any cause
Progression-free survival | 2 years
  Progression as determined by the clinician according to RECIST 1.1 definitions
Time to second line therapy | 2 years
  Date of starting sunitinib treatment to the date further systemic therapy is started

CONTACTS AND LOCATIONS:
Overall Officials: Howard Gurney, MBBS, FRACP, Principal Investigator — Crown Princess Mary Cancer Centre, Westmead
Locations (1):
- Crown Princess Mary Cancer Centre, Westmead Hospital, Westmead, New South Wales, Australia